CLINICAL TRIAL: NCT03557736
Title: Effects of a 12-Week Home-Based High-Intensity Interval Training Programme in Obese Individuals With Elevated Cardiovascular Disease Risk: A Pilot Study
Brief Title: Home-Based HIT in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Sam Shepherd, Dr Sam Shepherd, Liverpool John Moores University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Home-HIT
Record Dates: First submitted 2018-05-09; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Obese
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home-HIT (Experimental): Home-based high-intensity interval training: participants performed 12 weeks of simple body weight exercises in a place of their own choosing 3x/week
  Interventions: Behavioral: Training mode
- Home-MICT (Experimental): Home-based moderate-intensity interval training: participants performed 12 weeks of continuous exercise (running, swimming or cycling) in a place of their own choosing 3x/week
  Interventions: Behavioral: Training mode
- Lab-HIT (Experimental): Laboratory-based high-intensity interval training: participants performed supervised cycle exercise under laboratory conditions 3x/week for 12 weeks
  Interventions: Behavioral: Training mode

INTERVENTIONS:
Behavioral: Training mode — type of exercise training completed for 12 weeks

SUMMARY:
This study aims to investigate the efficacy of a novel home-based high-intensity interval training (Home-HIT) intervention in obese individuals, with elevated cardiovascular disease (CVD) risk. It was hypothesised that Home-HIT would 1) have high adherence to the prescribed exercise intensity (compliance), 2) improve markers of CVD risk, and 3) lead to favourable skeletal muscle adaptations.

DETAILED DESCRIPTION:
The applicability of current high intensity interval training (HIT) protocols to the sedentary obese population has been disputed by public health experts. Existing HIT interventions have been successful only under optimal conditions with high levels of supervision and specialised equipment, creating further barriers to exercise in those most in need. We aimed to eliminate many of these barriers by modifying existing HIT protocols to create a new home-based HIT (Home-HIT) intervention tailored to individuals with low fitness and mobility. It was hypothesised that Home-HIT would 1) have high adherence to the prescribed exercise intensity (compliance) and 2) improve markers of cardiovascular disease (CVD) risk. 32 Obese adults with at least 3 additional CVD risk factors (age 36±2 y; BMI 34.3±0.8 kg∙m-2; VO2peak 24.6±1.0 ml∙kg∙min-1), completed one of three 12-week training programmes 3x/week: Home-HIT (n=9); Laboratory-based supervised HIT (Lab-HIT; n=10) or home-based moderate intensity continuous training (Home-MICT; n=13). Adherence and compliance were monitored online in almost "real time" using a heart rate (HR) monitor and mobile app. The Home-HIT group completed 4 progressing to 8 1min intervals interspersed with 1min of rest in an unsupervised place of their choosing. The intervals were composed of simple bodyweight exercises that required no equipment. Changes in VO2peak, insulin sensitivity, body composition, flow-mediated dilation (FMD) and aortic pulse wave velocity (PWV) were assessed. Muscle biopsies were taken to assess changes in capillarisation, mitochondrial density, intramuscular triglyceride (IMTG) content and eNOS and GLUT4 protein expression using quantitative immunofluorescence microscopy.

ELIGIBILITY:
Inclusion Criteria:

* obesity (BMI >30 kg/m2)
* age 18-55

Exclusion Criteria:

* diagnosed CVD and other contraindications to participate in an exercise intervention
* BMI <30 kg/m2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
change in aerobic fitness | change in baseline aerobic fitness at 12 weeks
  change in maximal aerobic capacity following the training
Adherence and compliance to the exercise training intervention | adherance and compliance to the training over the 12 weeks
  Session completion rate (adherence) and ability to meet target heart rates (compliance)

SECONDARY OUTCOMES:
change in baseline FMD | change in baseline FMD at 12 weeks
  endothelial function measured using flow-mediated dilation (FMD)
change in vascular stiffness | change in baseline vascular stiffness at 12 weeks
  change in vascular stiffness with training
change in body fat percentage | chage in baseline body fat percentage at 12 weeks
  change in body fat percentage using DXA with training

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
there is no plan to share data with other researchers

REFERENCES:
- [Derived] Scott SN, Shepherd SO, Hopkins N, Dawson EA, Strauss JA, Wright DJ, Cooper RG, Kumar P, Wagenmakers AJM, Cocks M. Home-hit improves muscle capillarisation and eNOS/NAD(P)Hoxidase protein ratio in obese individuals with elevated cardiovascular disease risk. J Physiol. 2019 Aug;597(16):4203-4225. doi: 10.1113/JP278062. Epub 2019 Jul 15. PMID 31218680